CLINICAL TRIAL: NCT03689816
Title: The Impact of Bariatric Surgery on Estimated Bone Mineral Density in Chinese Obesity Patients: a Retrospective Cohort Study
Brief Title: the Related Factors of Bariatric Surgery on Bone Mineral Density
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, Jingge Yang, Director of bariatric surgery, First Affiliated Hospital of Jinan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstJinanU20180216
Record Dates: First submitted 2018-06-03; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Bone Mineral; Bariatric Surgery
MeSH Terms: interventions — Gastric Bypass

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bone density (Experimental): bone density
  Interventions: Procedure: sleeve gastrectomy; Procedure: gastric bypass

INTERVENTIONS:
Procedure: sleeve gastrectomy — sleeve gastrectomy
Procedure: gastric bypass — gastric bypass

SUMMARY:
Obesity and related metabolic diseases have become a chronic disease that is a threat to human health. Bariatric surgery can effectively and long-term reduce excess body weight and relieve related metabolic diseases, including type 2 diabetes. Laparoscopic gastric bypass surgery and laparoscopic sleeve gastrectomy are commonly used in bariatric surgery. Laparoscopic sleeve gastrectomy due to simple operation, good weight loss, and metabolic disease control effect, which is more widely used. However, there are several studies that show an increased chance of gastroesophageal reflux disease after laparoscopic sleeve gastrectomy. Long-term gastroesophageal reflux may lead to Barrett's esophagus or esophageal cancer. Nowadays, the cause of gastroesophageal reflux disease after sleeve gastrectomy is not clear and precautionary measures are not precise.

In this study, prospective randomized controlled trials were conducted to explore the possible causes of bone mineral after bariatric surgery and to explore ways to prevent bone mineral after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

-For the choice of surgical approach, numerous studies have shown that BMI ≧ 45, the general choice of gastric bypass surgery, BMI <45, you can choose sleeve gastrectomy. The remission rate for T2DM, sleeve gastrectomy has a good result for young patients with shorter duration. In our country, the BMI less than 45 is majorities.

Exclusion Criteria:

-BMI<27.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Preoperative of bone density | Preoperative
  bone density in g/cm3
Postoperative of bone density at 3 months | 3 months
  bone density in g/cm3
Postoperative of bone density at 6 months | 6 months
  bone density in g/cm3
Postoperative of bone density at 1 year | 1 year
  bone density in g/cm3

CONTACTS AND LOCATIONS:
Locations (1):
- The frist affiliated hospital of Jinan University, Guangzhou, Guangdong, China